CLINICAL TRIAL: NCT03847103
Title: Effects of Robotic-aided Therapy Combined With Bilateral Arm Training on Motor Performance and Electrophysiological Parameters of Upper Extremity for the Stroke Patients
Brief Title: Robotic-assisted Therapy With Bilateral Practice Improves Task and Motor Performance of the Upper Extremity for Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-ER-102-247
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Stroke Rehabilitation
Keywords: Stroke; Robotic-Assisted Therapy; Bilateral Practice; Task-specific Training; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic-aided rehabilitation with bilateral practice (Experimental): In addition to a 10-minutes sensorimotor stimulation programs, the experimental group received 40-minutes Robotic-assisted Therapy with Bilateral Practice programs.
  Interventions: Other: Robotic-assisted Therapy with Bilateral Practice; Other: Sensorimotor Stimulation Program
- Unilateral task-specific training (Active Comparator): In addition to a 10-minutes sensorimotor stimulation programs, the control subjects received 40-minute unilateral task-specific training.
  Interventions: Other: Unilateral Task-specific Training; Other: Sensorimotor Stimulation Program

INTERVENTIONS:
Other: Robotic-assisted Therapy with Bilateral Practice — 40-minute robotic-assisted therapy with bilateral practice program for wrist and forearm repetitive movement training was performed during each session.
  Arms: Robotic-aided rehabilitation with bilateral practice
Other: Unilateral Task-specific Training — 40 -minute unilateral task-specific training using various tasks: picks up beans with spoon, pouring water from one glass to another glass, opening and closing a drawer, drinking from a mug, and wiping the table were chosen for facilitating multitude of upper extremity functions. Three tasks per session were chosen for various specific components of hand-arm function training.
  Arms: Unilateral task-specific training
Other: Sensorimotor Stimulation Program — 10-minute sensorimotor stimulation program with repetitive range of motion exercises of upper extremity, proprioceptive neuromuscular facilitation and Rood approach

SUMMARY:
Task-specific repetitive training, an usual care in occupational therapy practice, and robotic-aided rehabilitation with bilateral practice to improve limb's movement control has been popularised; however the difference in treatment effects between this two therapeutic strategies has been rarely described. The aim of the study was to compare the efficacy of robotic-assisted therapy with bilateral practice (RTBP) and usual care on task and motor performance for chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke patients with unilateral cerebral infarction or hemorrhage and whose disease duration was more than six months following stroke
* no evidence of any other cerebral pathology in study screening CT scan
* a score for the Fugl-Meyer upper extremity motor assessment ranging from 23-53 corresponding to poor to notable arm-hand capacity
* pre stroke ability to speak the Chinese
* without any other possible somatic sensory impairment, no major cognitive-perceptual deficit based on the results of selective neuropsychological tests, such as the mini-mental state examination (MMSE) and Lowenstein occupational therapy cognitive assessment (LOTCA)
* premorbid right-handedness

Exclusion Criteria:

* less than six months following stroke
* CT shows multiple cerebral infarction or hemorrhage
* whose comprehension skills were insufficient to understand instructions
* individuals whose score of MMSE was lower than 24 or sub-item scores of visual perception, spatial perception, praxis, and visuomotor organization in LOTCA was lower than 8, 6, 6, and 14, respectively
* premorbid left-handedness

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Change in the result of Motor Activity Log | Baseline, endpoint (4 weeks) and follow-up (16 weeks) assessments
  Motor activity log is a structured interview with testing sensitivity used to examine how much (amount of use, AOU) and how well (quality of movement, QOM) the subject uses their more-affected arm. For the 30 items MAL, each item is scored on a 0-5-ordinal scale.

SECONDARY OUTCOMES:
Change in the result of Fugl-Meyer assessment for UE motor function | Baseline, endpoint (4 weeks) and follow-up (16 weeks) assessments
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.
Change in root mean square (RMS) value and the median frequency of the power spectrum of each detected motor unit action potential during maximum voluntary contraction | Baseline, endpoint (4 weeks) and follow-up (16 weeks) assessments
  Power and frequency function of Surface Electromyogram signals are reliable parameter to evaluate motor behavior of stroke survivors. The location sEMG electrodes were placed on the muscle belly of the anterior deltoid, flexor carpi radialis and extensor carpi radialis of the affected forearm.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Hsu HY, Chiu HY, Kuan TS, Tsai CL, Su FC, Kuo LC. Robotic-assisted therapy with bilateral practice improves task and motor performance in the upper extremities of chronic stroke patients: A randomised controlled trial. Aust Occup Ther J. 2019 Oct;66(5):637-647. doi: 10.1111/1440-1630.12602. Epub 2019 Jul 17. PMID 31317553